CLINICAL TRIAL: NCT00797927
Title: Quetiapine Related Neurochemical Changes as Measured by Magnetic Resonance Spectroscopy in Patients With Schizophrenia
Brief Title: Quetiapine Related Neurochemical Changes as Measured by Magnetic Resonance Spectroscopy in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Tzung-Jeng Hwang, attending psychiatrist, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200702010M
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; quetiapine; conventional antipsychotics; magnetic resonance spectroscopy
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. quetiapine (Experimental): quetiapine would replace the original conventional antipsychotic agent
  Interventions: Drug: quetiapine
- 2. conventional antipsychotics (No Intervention)
  Interventions: Other: no intervention

INTERVENTIONS:
Drug: quetiapine — quetiapine (with equivalent dose to original antipsychotic agent) would replace the original antipsychotic agent for 28 days
  Other Names: seroquel
  Arms: 1. quetiapine
Other: no intervention — keep the original conventional antipsychotic agent for 28 days
  Other Names: typical antipsychotics
  Arms: 2. conventional antipsychotics

SUMMARY:
we aim to examine whether a representative atypical antipsychotic, quetiapine, has different effects from conventional antipsychotics on the magnetic resonance spectroscopy (MRS) markers in schizophrenia patients.

DETAILED DESCRIPTION:
The impact of medications on MRS changes in brain of schizophrenia patients have rarely been studied through a well-controlled study. Most of the MRS studies in schizophrenia patients are cross-sectional and uncontrolled and devoid of any comparison between effects of different drugs. To date, only limited research has explored this issue and the results are conflicting. These conflicting results may be related to small sample size, different patient population and design in these studies. Thus, further studies are warranted. Besides, with the advent of new generation atypical antipsychotics, it will be important to know whether atypical antipsychotics exert different effects on neurons from conventional antipsychotics. If neuronal activity can be improved by atypical antipsychotics, the findings will have great clinical implications.

Fifteen patients in the experimental group will receive MRS examinations (including bilateral frontal and temporal area) in two phases: baseline (when they are on a conventional antipsychotic) and 4 weeks after shifting from that conventional antipsychotic to quetiapine. Another 15 schizophrenia patients receiving conventional antipsychotics will serve as the control group. The control group will receive the MRS examinations twice (baseline and 4 weeks later) without change of medications. In each phase, every patient will also receive the Positive and Negative Syndrome Scale (PANSS) assessment. The changes of the MRS markers will be analyzed and compared, both within and between the 2 groups, and their correlations with the PANSS scores will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. A diagnosis of schizophrenia or schizoaffective disorder by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
3. Females or males aged > 20 and < 65 years
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
5. Able to understand and comply with the requirements of the study
6. Undergoing treatment with a conventional antipsychotic drug and is clinically stable

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampicin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment as judged by the investigator
11. Involvement in the planning and conduct of the study
12. Previous enrolment or randomisation of treatment in the present study.
13. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
14. Subjects with metal prosthesis such as cardiac valves etc
15. Severe neurological co-morbidity such as stroke, encephalopathy etc or medical conditions that will compromise on the safety of patients such as acute myocardial infarction, systemic infections etc as judged by the investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The change from baseline in neurochemical peak area ratios (NAA/CRE, NAA/CHO, CHO/CRE) at the end of study | baseline and 28 th day

SECONDARY OUTCOMES:
changes from baseline in PANSS | baseline and 28th day

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Jeng Hwang, MD, Principal Investigator — Department of Psychiatry, National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan